CLINICAL TRIAL: NCT05712200
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to evaLuate the effIcacy and Safety of abeLacimab in High-risk Patients With Atrial Fibrillation Who Have Been Deemed Unsuitable for Oral antiCoagulation (LILAC-TIMI 76)
Brief Title: Study to evaLuate the effIcacy and Safety of abeLacimab in High-risk Patients With Atrial Fibrillation Who Have Been Deemed Unsuitable for Oral antiCoagulation (LILAC-TIMI 76)
Acronym: LILAC-TIMI 76
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anthos Therapeutics, Inc. (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANT-010; 2023-503224-66-00 (EU CTIS Number); CMAA868A2302 (Other: Novartis)
Record Dates: First submitted 2023-01-12; First posted 2023-02-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF)
Keywords: abelacimab; randomized; placebo-controlled; double-blind; endpoint evaluation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — abelacimab; MAA868

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abelacimab (MAA868) (Experimental): Patients will be randomized in a 1:1 ratio to receive abelacimab 150 mg subcutaneous (SC) or matching placebo once monthly.
  Interventions: Biological: Abelacimab
- Placebo (Placebo Comparator): Patients will be randomized in a 1:1 ratio to receive abelacimab 150 mg subcutaneous (SC) or matching placebo once monthly.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Abelacimab — Abelacimab provided as liquid in vial (150 mg/mL)
  Other Names: MAA868
  Arms: Abelacimab (MAA868)
Drug: Placebo — Dosage Formulation: Liquid (in vial)
  Dose Strength: Placebo to Abelacimab
  Arms: Placebo

SUMMARY:
A study to evaluate the effect of abelacimab relative to placebo on the rate of ischemic stroke or systemic embolism (SE) in patients with Atrial Fibrillation (AF) who have been deemed by their responsible physicians or by their own decision to be unsuitable for oral anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to understand and has provided written informed consent to participate in the trial
* Diagnosed Atrial Fibrillation (AF) or atrial flutter (documented on an electrocardiogram (ECG) or monitor recording)
* Age 65-74 and a CHA2DS2VASc ≥4 OR age ≥75 and a CHA2DS2VASc ≥3
* Patient is judged by the responsible physician to be unsuitable for oral anticoagulation because the risks outweigh the benefits or the patient is unwilling to take oral anticoagulation AND this determination was made prior to and independent of the study
* At least 1 bleeding risk factor such as severe renal insufficiency, planned daily use of antiplatelet medication for the duration of the trial, history of bleeding from a critical area, or other conditions associated with increased risk of bleeding such as chronic nonsteroidal anti-inflammatory drug (NSAID) use, frailty or multiple falls
* Patient is judged by the responsible physician to be unsuitable for left atrial appendage (LAA) closure or occlusion device, an approved device is not available, or the patient is unwilling to undergo the procedure AND this determination was made prior to and independent of the study

Exclusion Criteria:

* AF due to an ongoing acute reversible cause (e.g., cardiac surgery, pulmonary embolism (PE), untreated hyperthyroidism, alcohol use)
* Patients who within 60 days prior to randomization (1) received a vitamin K antagonists (VKA) (e.g., warfarin, phenprocoumon, acenocoumarol) or a direct oral anticoagulant (DOAC) such as, dabigatran, rivaroxaban, apixaban, or edoxaban or (2) were newly diagnosed with AF
* Patients with an intracranial or intraocular bleed within the 3 months prior to screening or any history of spontaneous intracerebral hemorrhage at any time in the absence of antithrombotic treatment
* Any stroke within 14 days before randomization or transient ischemic attack (TIA) within 3 days before randomization
* Mechanical heart valve or valve disease that is expected to require mechanical valve replacement intervention (surgical or invasive) during the course of the study
* Patients on dialysis at screening or who are planned to start dialysis within 6 months

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Time to first event of ischemic stroke or systemic embolism (SE) | Up to 30 months
Safety: Time to first occurrence of Bleeding Academic Research Consortium (BARC) type 3c/5 bleeding | Up to 30 months

SECONDARY OUTCOMES:
Efficacy: Time to first event of ischemic stroke, systemic embolism (SE), myocardial infarctions (MI), venous thromboembolism (VTE), or acute limb ischemia | Up to 30 months
  Abelacimab versus placebo with regard to the composite of ischemic stroke, SE, MI, VTE, or acute limb ischemia
Efficacy: Time to first event of ischemic stroke, systemic embolism (SE), or Bleeding Academic Research Consortium (BARC) type 3c/5 bleeding event | Up to 30 months
Efficacy: Cardiovascular (CV) mortality | Up to 30 months
Efficacy: All-cause mortality | Up to 30 months
Time to first event of ischemic stroke, systemic embolism (SE), myocardial infarctions (MI), venous thromboembolism (VTE), acute limb ischemia, or International Society on Thrombosis and Haemostasis (ISTH) major bleeding | Up to 30 months
  Abelacimab versus placebo with regard to net clinical outcome defined as the composite of ischemic stroke, SE, MI, VTE, acute limb ischemia, or International Society on Thrombosis and Haemostasis (ISTH) major bleeding

CONTACTS AND LOCATIONS:
Locations (681):
- United States (140):
  - Anthos Investigative Site 1040, Birmingham, Alabama
  - Anthos Investigative Site 9947, Birmingham, Alabama
  - Anthos Investigative Site 1041, Mobile, Alabama
  - Anthos Investigative Site 1089, Gilbert, Arizona
  - Anthos Investigative Site 1099, Peoria, Arizona
  - Anthos Investigative Site 9906, Phoenix, Arizona
  - Anthos Investigative Site 9927, Yuma, Arizona
  - Anthos Investigative Site 9929, Huntington Beach, California
  - Anthos Investigative Site 9959, Imperial, California
  - Anthos Investigative Site 9921, Lancaster, California
  - Anthos Investigative Site 1078, Loma Linda, California
  - Anthos Investigative Site 1077, Los Angeles, California
  - Anthos Investigative Site 1015, Northridge, California
  - Anthos Investigative Site 1070, Redding, California
  - Anthos Investigative Site 1071, San Dimas, California
  - Anthos Investigative Site 1076, Santa Ana, California
  - Anthos Investigative Site 9938, Santa Rosa, California
  - Anthos Investigative Site 9908, South Gate, California
  - Anthos Investigative Site 9907, Vista, California
  - Anthos Investigative Site 1095, Aurora, Colorado
  - Anthos Investigative Site 1049, Denver, Colorado
  - Anthos Investigative Site 9922, Golden, Colorado
  - Anthos Investigative Site 1012, Stamford, Connecticut
  - Anthos Investigative Site 9934, Altamonte Springs, Florida
  - Anthos Investigative Site 1013, Boca Raton, Florida
  - Anthos Investigative Site 1025, Clearwater, Florida
  - Anthos Investigative Site 1022, Clearwater, Florida
  - Anthos Investigative Site 1019, Daytona Beach, Florida
  - Anthos Investigative Site 9936, Hialeah, Florida
  - Anthos Investigative Site 1083, Hollywood, Florida
  - Anthos Investigative Site 1008, Jacksonville, Florida
  - Anthos Investigative Site 9904, Lake Mary, Florida
  - Anthos Investigative Site 1093, Lutz, Florida
  - Anthos Investigative Site 9933, Miami, Florida
  - Anthos Investigative Site 1072, Miami Lakes, Florida
  - Anthos Investigative Site 9944, Ocala, Florida
  - Anthos Investigative Site 9940, Ocala, Florida
  - Anthos Investigative Site 1067, Ormond Beach, Florida
  - Anthos Investigative Site 1026, Safety Harbor, Florida
  - Anthos Investigative Site 1002, Saint Augustine, Florida
  - Anthos Investigative Site 1004, Saint Augustine, Florida
  - Anthos Investigative Site 1044, Tamarac, Florida
  - Anthos Investigative Site 1088, Tamarac, Florida
  - Anthos Investigative Site 1046, Tampa, Florida
  - Anthos Investigative Site 9911, The Villages, Florida
  - Anthos Investigative Site 1052, Lithonia, Georgia
  - Anthos Investigative Site 1033, Macon, Georgia
  - Anthos Investigative Site 1042, Norcross, Georgia
  - Anthos Investigative Site 1003, Suwanee, Georgia
  - Anthos Investigative Site 9953, Tucker, Georgia
  - Anthos Investigative Site 1030, Park Ridge, Illinois
  - Anthos Investigative Site 9932, Rockford, Illinois
  - Anthos Investigative Site 9925, Winfield, Illinois
  - Anthos Investigative Site 9915, Evansville, Indiana
  - Anthos Investigative Site 1098, Merrillville, Indiana
  - Anthos Investigative Site 9956, West Des Moines, Iowa
  - Anthos Investigative Site 9958, Hutchinson, Kansas
  - Anthos Investigative Site 1016, Wichita, Kansas
  - Anthos Investigative Site 1006, Alexandria, Louisiana
  - Anthos Investigative Site 1043, Shreveport, Louisiana
  - Anthos Investigative Site 1054, Bangor, Maine
  - Anthos Investigative Site 1039, Baltimore, Maryland
  - Anthos Investigative Site 1023, Lanham, Maryland
  - Anthos Investigative Site 1028, Rockville, Maryland
  - Anthos Investigative Site 1082, Boston, Massachusetts
  - Anthos Investigative Site 9918, Boston, Massachusetts
  - Anthos Investigative Site 1021, Lansing, Michigan
  - Anthos Investigative Site 9946, Petoskey, Michigan
  - Anthos Investigative Site 1059, Southgate, Michigan
  - Anthos Investigative Site 1017, Tupelo, Mississippi
  - Anthos Investigative Site 1080, Kansa City, Missouri
  - Anthos Investigative Site 9948, Kansas City, Missouri
  - Anthos Investigative Site 1066, Lincoln, Nebraska
  - Anthos Investigative Site 1036, Las Vegas, Nevada
  - Anthos Investigative Site 9914, Las Vegas, Nevada
  - Anthos Investigative Site 1094, Englewood, New Jersey
  - Anthos Investigative Site 9931, Albany, New York
  - Anthos Investigative Site 9905, Brooklyn, New York
  - Anthos Investigative Site 1014, Middletown, New York
  - Anthos Investigative Site 1037, Rosedale, New York
  - Anthos Investigative Site 9935, Stony Brook, New York
  - Anthos Investigative Site 9920, Valhalla, New York
  - Anthos Investigative Site 9924, Westfield, New York
  - Anthos Investigative Site 1065, Cary, North Carolina
  - Anthos Investigative Site 1005, Charlotte, North Carolina
  - Anthos Investigative Site 9912, Durham, North Carolina
  - Anthos Investigative Site 1048, Fayetteville, North Carolina
  - Anthos Investigative Site 1035, Henderson, North Carolina
  - Anthos Investigative Site 1001, Lenoir, North Carolina
  - Anthos Investigative Site 9950, Pinehurst, North Carolina
  - Anthos Investigative Site 9951, Statesville, North Carolina
  - Anthos Investigative Site 9952, Wilmington, North Carolina
  - Anthos Investigative Site 9902, Beavercreek, Ohio
  - Anthos Investigative Site 9945, Dayton, Ohio
  - Anthos Investigative Site 9917, Oklahoma City, Oklahoma
  - Anthos Investigative Site 1075, Portland, Oregon
  - Anthos Investigative Site 1074, Bristol, Pennsylvania
  - Anthos Investigative Site 1087, Horsham, Pennsylvania
  - Anthos Investigative Site 1032, Rock Hill, South Carolina
  - Anthos Investigative Site 1050, Elizabethton, Tennessee
  - Anthos Investigative Site 1057, Germantown, Tennessee
  - Anthos Investigative Site 9941, Jefferson City, Tennessee
  - Anthos Investigative Site 1056, Memphis, Tennessee
  - Anthos Investigative Site 9928, Allen, Texas
  - Anthos Investigative Site 9913, Beaumont, Texas
  - Anthos Investigative Site 9943, Dallas, Texas
  - Anthos Investigative Site 9942, Dallas, Texas
  - Anthos Investigative Site 1091, El Paso, Texas
  - Anthos Investigative Site 9930, Greenville, Texas
  - Anthos Investigative Site 1069, Houston, Texas
  - Anthos Investigative Site 1068, Houston, Texas
  - Anthos Investigative Site 1097, Houston, Texas
  - Anthos Investigative Site 9903, Houston, Texas
  - Anthos Investigative Site 1053, Houston, Texas
  - Anthos Investigative Site 1064, Houston, Texas
  - Anthos Investigative Site 9901, Laredo, Texas
  - Anthos Investigative Site 1063, McAllen, Texas
  - Anthos Investigative Site 1096, McKinney, Texas
  - Anthos Investigative Site 1079, McKinney, Texas
  - Anthos Investigative Site 1024, Odessa, Texas
  - Anthos Investigative Site 1085, Port Arthur, Texas
  - Anthos Investigative Site 9923, Sherman, Texas
  - Anthos Investigative Site 1090, Sugar Land, Texas
  - Anthos Investigative Site 1011, Tomball, Texas
  - Anthos Investigative Site 9916, Tyler, Texas
  - Anthos Investigative Site 9910, Victoria, Texas
  - Anthos Investigative Site 1060, Waco, Texas
  - Anthos Investigative Site 9909, Webster, Texas
  - Anthos Investigative Site 1092, Wylie, Texas
  - Anthos Investigative Site 1084, American Fork, Utah
  - Anthos Investigative Site 1031, Bountiful, Utah
  - Anthos Investigative Site 1029, Holladay, Utah
  - Anthos Investigative Site 1038, Pleasant View, Utah
  - Anthos Investigative Site 1034, Roy, Utah
  - Anthos Investigative Site 1018, Falls Church, Virginia
  - Anthos Investigative Site 1010, Manassas, Virginia
  - Anthos Investigative Site 1009, Roanoke, Virginia
  - Anthos Investigative Site 9949, Vienna, Virginia
  - Anthos Investigative Site 9926, Redmond, Washington
  - Anthos Investigative Site 1073, Tacoma, Washington
- Argentina (24):
  - Anthos Investigative Site 1411, Buenos Aires
  - Anthos Investigative Site 1430, Buenos Aires
  - Anthos Investigative Site 1409, Ciudad Autónoma Buenos Aires
  - Anthos Investigative Site 1410, Ciudad Autónoma de Buenos Aire
  - Anthos Investigative Site 1423, Ciudad Autónoma de Buenos Aire
  - Anthos Investigative Site 1429, Coronel Suárez
  - Anthos Investigative Site 1420, Corrientes
  - Anthos Investigative Site 1407, Córdoba
  - Anthos Investigative Site 1414, Córdoba
  - Anthos Investigative Site 1418, Córdoba
  - Anthos Investigative Site 1424, Córdoba
  - Anthos Investigative Site 1427, Córdoba
  - Anthos Investigative Site 1434, Córdoba
  - Anthos Investigative Site 1419, Córdoba
  - Anthos Investigative Site 1431, Córdoba
  - Anthos Investigative Site 1402, La Plata
  - Anthos Investigative Site 1417, Quilmes
  - Anthos Investigative Site 1415, Ramos Mejía
  - Anthos Investigative Site 1403, Salta
  - Anthos Investigative Site 1425, San Luis
  - Anthos Investigative Site 1426, San Martín
  - Anthos Investigative Site 1404, San Miguel de Tucumán
  - Anthos Investigative Site 1435, San Miguel de Tucumán
  - Anthos Investigative Site 1436, San Nicolás
- Brazil (43):
  - Anthos Investigative Site 1518, Aracaju
  - Anthos Investigative Site 1527, Belo Horizonte
  - Anthos Investigative Site 1528, Belo Horizonte
  - Anthos Investigative Site 1516, Belo Horizonte
  - Anthos Investigative Site 1507, Belo Horizonte
  - Anthos Investigative Site 1513, Blumenau
  - Anthos Investigative Site 1505, Blumenau
  - Anthos Investigative Site 1535, Brasília
  - Anthos Investigative Site 1501, Campina Grande do Sul
  - Anthos Investigative Site 1503, Campinas
  - Anthos Investigative Site 1522, Campinas
  - Anthos Investigative Site 1520, Campo Grande
  - Anthos Investigative Site 1532, Canoas
  - Anthos Investigative Site 1526, Caxias do Sul
  - Anthos Investigative Site 1542, Colatina
  - Anthos Investigative Site 1540, Curitiba
  - Anthos Investigative Site 1509, Curitiba
  - Anthos Investigative Site 1525, Goiânia
  - Anthos Investigative Site 1502, Marília
  - Anthos Investigative Site 1533, Passo Fundo
  - Anthos Investigative Site 1517, Porto Alegre
  - Anthos Investigative Site 1519, Porto Alegre
  - Anthos Investigative Site 1544, Porto Alegre
  - Anthos Investigative Site 1506, Porto Alegre
  - Anthos Investigative Site 1530, Porto Alegre
  - Anthos Investigative Site 1512, Porto Alegre
  - Anthos Investigative Site 1524, Porto Alegre
  - Anthos Investigative Site 1508, Porto Alegre
  - Anthos Investigative Site 1531, Recife
  - Anthos Investigative Site 1515, Ribeirão Preto
  - Anthos Investigative Site 1536, Ribeirão Preto
  - Anthos Investigative Site 1537, Rio de Janeiro
  - Anthos Investigative Site 1510, Salvador
  - Anthos Investigative Site 1521, Salvador
  - Anthos Investigative Site 1534, São Paulo
  - Anthos Investigative Site 1511, São Paulo
  - Anthos Investigative Site 1538, São Paulo
  - Anthos Investigative Site 1539, São Paulo
  - Anthos Investigative Site 1529, São Paulo
  - Anthos Investigative Site 1543, São Paulo
  - Anthos Investigative Site 1514, Tatuí
  - Anthos Investigative Site 1541, Teresina
  - Anthos Investigative Site 1504, Votuporanga
- Bulgaria (31):
  - Anthos Investigative Site 6014, Blagoevgrad
  - Anthos Investigative Site 6026, Burgas
  - Anthos Investigative Site 6019, Gabrovo
  - Anthos Investigative Site 6032, Haskovo
  - Anthos Investigative Site 6018, Haskovo
  - Anthos Investigative Site 6013, Panagyurishte
  - Anthos Investigative Site 6025, Pazardzhik
  - Anthos Investigative Site 6006, Pleven
  - Anthos Investigative Site 6003, Pleven
  - Anthos Investigative Site 6007, Plovdiv
  - Anthos Investigative Site 6008, Plovdiv
  - Anthos Investigative Site 6009, Plovdiv
  - Anthos Investigative Site 6004, Plovdiv
  - Anthos Investigative Site 6021, Plovdiv
  - Anthos Investigative Site 6031, Rousse
  - Anthos Investigative Site 6027, Sliven
  - Anthos Investigative Site 6034, Sliven
  - Anthos Investigative Site 6022, Smolyan
  - Anthos Investigative Site 6030, Sofia
  - Anthos Investigative Site 6028, Sofia
  - Anthos Investigative Site 6029, Sofia
  - Anthos Investigative Site 6024, Sofia
  - Anthos Investigative Site 6023, Sofia
  - Anthos Investigative Site 6010, Sofia
  - Anthos Investigative Site 6015, Sofia
  - Anthos Investigative Site 6020, Sofia
  - Anthos Investigative Site 6001, Sofia
  - Anthos Investigative Site 6017, Sofia
  - Anthos Investigative Site 6012, Sofia
  - Anthos Investigative Site 6002, Sofia
  - Anthos Investigative Site 6011, Stara Zagora
- Canada (23):
  - Anthos Investigative Site 2012, Mira Road, Nova Scotia
  - Anthos Investigative Site 2003, Cambridge, Ontario
  - Anthos Investigative Site 2007, Chicoutimi, Quebec
  - Anthos Investigative Site 2010, Sherbrooke, Quebec
  - Anthos Investigative Site 2016, Abbotsford
  - Anthos Investigative Site 2019, Brampton
  - Anthos Investigative Site 2015, Edmonton
  - Anthos Investigative Site 2018, Greenfield Park
  - Anthos Investigative Site 2005, Halifax
  - Anthos Investigative Site 2025, Hamilton
  - Anthos Investigative Site 2026, Hamilton
  - Anthos Investigative Site 2028, Markham
  - Anthos Investigative Site 2014, Montreal
  - Anthos Investigative Site 2004, New Westminster
  - Anthos Investigative Site 2021, North Vancouver
  - Anthos Investigative Site 2002, Québec
  - Anthos Investigative Site 2024, Saint Catharines
  - Anthos Investigative Site 2006, Saint-Jérôme
  - Anthos Investigative Site 2027, Terrebonne
  - Anthos Investigative Site 2022, Thunder Bay
  - Anthos Investigative Site 2017, Toronto
  - Anthos Investigative Site 2020, Toronto
  - Anthos Investigative Site 2023, Toronto
- Chile (10):
  - Anthos Investigative Site 1605, Concepción
  - Anthos Investigative Site 1606, Independencia
  - Anthos Investigative Site 1604, Providencia
  - Anthos Investigative Site 1607, San Bernardo
  - Anthos Investigative Site 1609, San Miguel
  - Anthos Investigative Site 1608, Santiago
  - Anthos Investigative Site 1610, Talcahuano
  - Anthos Investigative Site 1603, Temuco
  - Anthos Investigative Site 1602, Temuco
  - Anthos Investigative Site 1601, Viña del Mar
- China (22):
  - Anthos Investigative Site 1834, Shantou, Guangdong
  - Anthos Investigative Site 1837, Wuhan, Hubei
  - Anthos Investigative Site 1821, Xi'an, Shaanxi
  - Anthos Investigative Site 1818, Changchun
  - Anthos Investigative Site 1810, Changsha
  - Anthos Investigative Site 1811, Changsha
  - Anthos Investigative Site 1802, Chengdu
  - Anthos Investigative Site 1829, Guangzhou
  - Anthos Investigative Site 1809, Haidian
  - Anthos Investigative Site 1801, Hangzhou
  - Anthos Investigative Site 1808, Hangzhou
  - Anthos Investigative Site 1816, Jinan
  - Anthos Investigative Site 1804, Lianyungang
  - Anthos Investigative Site 1814, Luoyang
  - Anthos Investigative Site 1817, Nanchang
  - Anthos Investigative Site 1820, Nanchang
  - Anthos Investigative Site 1803, Nanjing
  - Anthos Investigative Site 1815, Ningbo
  - Anthos Investigative Site 1819, Shijiazhuang
  - Anthos Investigative Site 1812, Tianjin
  - Anthos Investigative Site 1813, Yangzhou
  - Anthos Investigative Site 1805, Yinchuan
- Colombia (12):
  - Anthos Investigative Site 2501, Manizales, Caldas Department
  - Anthos Investigative Site 2503, Armenia, QUI
  - Anthos Investigative Site 2513, Barranquilla
  - Anthos Investigative Site 2504, Barranquilla
  - Anthos Investigative Site 2512, Barranquilla
  - Anthos Investigative Site 2511, Cali
  - Anthos Investigative Site 2507, Cartagena
  - Anthos Investigative Site 2506, Floridablanca
  - Anthos Investigative Site 2508, Medellín
  - Anthos Investigative Site 2502, Pereira
  - Anthos Investigative Site 2510, Piedecuesta
  - Anthos Investigative Site 2505, Soledad
- Croatia (9):
  - Anthos Investigative Site 3102, Krapinske Toplice
  - Anthos Investigative Site 3108, Osijek
  - Anthos Investigative Site 3107, Rijeka
  - Anthos Investigative Site 3111, Zabok
  - Anthos Investigative Site 3109, Zadar
  - Anthos Investigative Site 3101, Zagreb
  - Anthos Investigative Site 3103, Zagreb
  - Anthos Investigative Site 3104, Zagreb
  - Anthos Investigative Site 3110, Zagreb
- Czechia (10):
  - Anthos Investigative Site 3002, Brandýs nad Labem
  - Anthos Investigative Site 3006, Liberec
  - Anthos Investigative Site 3007, Ostrava - Poruba
  - Anthos Investigative Site 3001, Poděbrady
  - Anthos Investigative Site 3005, Prague
  - Anthos Investigative Site 3004, Prague
  - Anthos Investigative Site 3003, Prague
  - Anthos Investigative Site 3010, Prague
  - Anthos Investigative Site 3009, Trutnov
  - Anthos Investigative Site 3011, Ústí nad Labem
- Estonia (3):
  - Anthos Investigative Site 2203, Tallinn
  - Anthos Investigative Site 2202, Tallinn
  - Anthos Investigative Site 2201, Tallinn
- Finland (2):
  - Anthos Investigative Site 3401, Joensuu
  - Anthos Investigative Site 3403, Turku
- Germany (10):
  - Anthos Investigative Site 7006, Altenburg
  - Anthos Investigative Site 7014, Berlin
  - Anthos Investigative Site 7004, Dresden
  - Anthos Investigative Site 7012, Hamburg
  - Anthos Investigative Site 7003, Hamburg
  - Anthos Investigative Site 7013, Hanover
  - Anthos Investigative Site 7009, Ludwigshafen
  - Anthos Investigative Site 7002, Markkleeberg
  - Anthos Investigative Site 7007, Paderborn
  - Anthos Investigative Site 7001, Schwerin
- Greece (11):
  - Anthos Investigative Site 2714, Athens
  - Anthos Investigative Site 2711, Athens
  - Anthos Investigative Site 2704, Athens
  - Anthos Investigative Site 2702, Cholargós
  - Anthos Investigative Site 2705, Glyfada
  - Anthos Investigative Site 2706, Larissa
  - Anthos Investigative Site 2712, Marousi
  - Anthos Investigative Site 2715, Rio
  - Anthos Investigative Site 2709, Thessaloniki
  - Anthos Investigative Site 2708, Thessaloniki
  - Anthos Investigative Site 2710, Voula
- Hungary (14):
  - Anthos Investigative Site 4002, Békéscsaba
  - Anthos Investigative Site 4015, Budapest
  - Anthos Investigative Site 4006, Budapest
  - Anthos Investigative Site 4009, Budapest
  - Anthos Investigative Site 4018, Budapest
  - Anthos Investigative Site 4014, Budapest
  - Anthos Investigative Site 4011, Gyöngyös
  - Anthos Investigative Site 4012, Kaposvár
  - Anthos Investigative Site 4007, Kistarcsa
  - Anthos Investigative Site 4005, Nyíregyháza
  - Anthos Investigative Site 4010, Pécs
  - Anthos Investigative Site 4017, Szeged
  - Anthos Investigative Site 4016, Veszprém
  - Anthos Investigative Site 4008, Zalaegerszeg
- India (34):
  - Anthos Investigative Site 2340, Kochi, Kerala
  - Anthos Investigative Site 2310, Ahmedabad
  - Anthos Investigative Site 2320, Ahmedabad
  - Anthos Investigative Site 2330, Ajmer
  - Anthos Investigative Site 2311, Bangalore
  - Anthos Investigative Site 2318, Bhubaneswar
  - Anthos Investigative Site 2303, Chandigarh
  - Anthos Investigative Site 2324, Chennai
  - Anthos Investigative Site 2338, Chennai
  - Anthos Investigative Site 2325, Chennai
  - Anthos Investigative Site 2328, Dehradun
  - Anthos Investigative Site 2308, Ghaziabad
  - Anthos Investigative Site 2333, Hyderabad
  - Anthos Investigative Site 2306, Jaipur
  - Anthos Investigative Site 2331, Jaipur
  - Anthos Investigative Site 2304, Kochi
  - Anthos Investigative Site 2314, Kolkata
  - Anthos Investigative Site 2323, Ludhiāna
  - Anthos Investigative Site 2326, Mangaluru
  - Anthos Investigative Site 2329, Meerut
  - Anthos Investigative Site 2313, Mumbai
  - Anthos Investigative Site 2315, Nagpur
  - Anthos Investigative Site 2336, Nagpur
  - Anthos Investigative Site 2316, Nagpur
  - Anthos Investigative Site 2307, New Delhi
  - Anthos Investigative Site 2301, New Delhi
  - Anthos Investigative Site 2319, New Delhi
  - Anthos Investigative Site 2327, New Delhi
  - Anthos Investigative Site 2322, New Delhi
  - Anthos Investigative Site 2305, Pune
  - Anthos Investigative Site 2317, Pune
  - Anthos Investigative Site 2309, Secunderabad
  - Anthos Investigative Site 2312, Visakhapatnam
  - Anthos Investigative Site 2321, Visakhapatnam
- Israel (13):
  - Anthos Investigative Site 1210, Afula
  - Anthos Investigative Site 1205, Ashkelon
  - Anthos Investigative Site 1213, Beersheba
  - Anthos Investigative Site 1206, Hadera
  - Anthos Investigative Site 1211, Haifa
  - Anthos Investigative Site 1201, Haifa
  - Anthos Investigative Site 1209, Holon
  - Anthos Investigative Site 1212, Jerusalem
  - Anthos Investigative Site 1204, Kfar Saba
  - Anthos Investigative Site 1202, Nahariya
  - Anthos Investigative Site 1207, Petah Tikva
  - Anthos Investigative Site 1203, Rehovot
  - Anthos Investigative Site 1208, Safed
- Italy (28):
  - Anthos Investigative Site 8016, Ancona
  - Anthos Investigative Site 8003, Bologna
  - Anthos Investigative Site 8015, Brescia
  - Anthos Investigative Site 8020, Cagliari
  - Anthos Investigative Site 8019, Caserta
  - Anthos Investigative Site 8008, Catanzaro
  - Anthos Investigative Site 8021, Cinisello Balsamo
  - Anthos Investigative Site 8024, Florence
  - Anthos Investigative Site 8013, Lecco
  - Anthos Investigative Site 8007, Milan
  - Anthos Investigative Site 8001, Milan
  - Anthos Investigative Site 8026, Naples
  - Anthos Investigative Site 8023, Napoli
  - Anthos Investigative Site 8017, Palermo
  - Anthos Investigative Site 8025, Pisa
  - Anthos Investigative Site 8029, Pisa
  - Anthos Investigative Site 8031, Ravenna
  - Anthos Investigative Site 8030, Rimini
  - Anthos Investigative Site 8028, Rivoli
  - Anthos Investigative Site 8010, Roma
  - Anthos Investigative Site 8011, Roma
  - Anthos Investigative Site 8002, Roma
  - Anthos Investigative Site 8022, Rome
  - Anthos Investigative Site 8004, Saronno
  - Anthos Investigative Site 8005, Sesto San Giovanni
  - Anthos Investigative Site 8014, Torino
  - Anthos Investigative Site 8006, Varese
  - Anthos Investigative Site 8009, Vittoria
- Japan (33):
  - Anthos Investigative Site 1923, Akashi
  - Anthos Investigative Site 1908, Chikushino-shi
  - Anthos Investigative Site 1902, Chūōku
  - Anthos Investigative Site 1920, Funabashi-Shi
  - Anthos Investigative Site 1910, Hamada-shi
  - Anthos Investigative Site 1924, Hamamatsu
  - Anthos Investigative Site 1906, Himeji-Shi
  - Anthos Investigative Site 1911, Imabari
  - Anthos Investigative Site 1912, Isehara-Shi
  - Anthos Investigative Site 1921, Kōtoku
  - Anthos Investigative Site 1915, Kure-shi
  - Anthos Investigative Site 1931, Matsue
  - Anthos Investigative Site 1903, Matsumoto-Shi
  - Anthos Investigative Site 1907, Nagano
  - Anthos Investigative Site 1929, Naha
  - Anthos Investigative Site 1934, Okayama
  - Anthos Investigative Site 1932, Osaka
  - Anthos Investigative Site 1930, Osaka
  - Anthos Investigative Site 1926, Ōmihachiman
  - Anthos Investigative Site 1922, Sapporo
  - Anthos Investigative Site 1904, Sendai
  - Anthos Investigative Site 1913, Shimonoseki-shi
  - Anthos Investigative Site 1914, Tachikawa-shi
  - Anthos Investigative Site 1909, Tochigi
  - Anthos Investigative Site 1925, Tokushima
  - Anthos Investigative Site 1933, Tokyo
  - Anthos Investigative Site 1928, Toyama
  - Anthos Investigative Site 1927, Tōon
  - Anthos Investigative Site 1901, Urayasu
  - Anthos Investigative Site 1917, Uwajima-Shi
  - Anthos Investigative Site 1918, Yokohama
  - Anthos Investigative Site 1919, Yokohama
  - Anthos Investigative Site 1916, Yokohama
- Latvia (11):
  - Anthos Investigative Site 2103, Baldone
  - Anthos Investigative Site 2109, Balvi
  - Anthos Investigative Site 2107, Daugavpils
  - Anthos Investigative Site 2108, Limbaži
  - Anthos Investigative Site 2110, Riga
  - Anthos Investigative Site 2101, Riga
  - Anthos Investigative Site 2105, Riga
  - Anthos Investigative Site 2102, Riga
  - Anthos Investigative Site 2111, Sigulda
  - Anthos Investigative Site 2104, Valmiera
  - Anthos Investigative Site 2106, Valmiera
- Malaysia (13):
  - Anthos Investigative Site 3513, Alor Star
  - Anthos Investigative Site 3501, Kajang
  - Anthos Investigative Site 3505, Kuala Lumpur
  - Anthos Investigative Site 3508, Kuantan
  - Anthos Investigative Site 3511, Kuantan
  - Anthos Investigative Site 3510, Kuching
  - Anthos Investigative Site 3503, Kuching
  - Anthos Investigative Site 3506, Miri
  - Anthos Investigative Site 3509, Putrajaya
  - Anthos Investigative Site 3502, Seberang Jaya
  - Anthos Investigative Site 3507, Seremban
  - Anthos Investigative Site 3512, Sibu
  - Anthos Investigative Site 3504, Sungai Buloh
- Mexico (17):
  - Anthos Investigative Site 1701, Aguascalientes
  - Anthos Investigative Site 1707, Aguascalientes
  - Anthos Investigative Site 1713, Aguascalientes
  - Anthos Investigative Site 1721, Chihuahua City
  - Anthos Investigative Site 1703, Culiacán
  - Anthos Investigative Site 1715, Guadalajara
  - Anthos Investigative Site 1711, Guerrero
  - Anthos Investigative Site 1712, Mexico City
  - Anthos Investigative Site 1704, Monterrey
  - Anthos Investigative Site 1705, Monterrey
  - Anthos Investigative Site 1719, Monterrey
  - Anthos Investigative Site 1702, Querétaro
  - Anthos Investigative Site 1718, San Luis Potosí City
  - Anthos Investigative Site 1716, Tlalpan
  - Anthos Investigative Site 1706, Veracruz
  - Anthos Investigative Site 1708, Veracruz
  - Anthos Investigative Site 1709, Xalapa
- Peru (3):
  - Anthos Investigative Site 3703, San Isidro, Lima region
  - Anthos Investigative Site 3706, Piura
  - Anthos Investigative Site 3708, San Borja
- Philippines (5):
  - Anthos Investigative Site 3603, Angeles City
  - Anthos Investigative Site 3601, Davao City
  - Anthos Investigative Site 3608, Iloilo City
  - Anthos Investigative Site 3610, Lahug
  - Anthos Investigative Site 3604, Lipa City
- Poland (32):
  - Anthos Investigative Site 5029, Bialystok
  - Anthos Investigative Site 5022, Czeladź
  - Anthos Investigative Site 5033, Elblag
  - Anthos Investigative Site 5010, Gdynia
  - Anthos Investigative Site 5034, Gdynia
  - Anthos Investigative Site 5003, Katowice
  - Anthos Investigative Site 5009, Katowice
  - Anthos Investigative Site 5030, Katowice
  - Anthos Investigative Site 5005, Katowice
  - Anthos Investigative Site 5016, Krakow
  - Anthos Investigative Site 5018, Krakow
  - Anthos Investigative Site 5032, Legnica
  - Anthos Investigative Site 5021, Lodz
  - Anthos Investigative Site 5012, Lodz
  - Anthos Investigative Site 5028, Lodz
  - Anthos Investigative Site 5023, Lublin
  - Anthos Investigative Site 5006, Lublin
  - Anthos Investigative Site 5039, Mielec
  - Anthos Investigative Site 5041, Nowa Sól
  - Anthos Investigative Site 5008, Olsztyn
  - Anthos Investigative Site 5025, Oświęcim
  - Anthos Investigative Site 5002, Przemyśl
  - Anthos Investigative Site 5004, Rzeszów
  - Anthos Investigative Site 5001, Tychy
  - Anthos Investigative Site 5014, Warsaw
  - Anthos Investigative Site 5038, Warsaw
  - Anthos Investigative Site 5017, Warsaw
  - Anthos Investigative Site 5011, Warsaw
  - Anthos Investigative Site 5015, Warsaw
  - Anthos Investigative Site 5019, Wroclaw
  - Anthos Investigative Site 5007, Wroclaw
  - Anthos Investigative Site 5024, Zabrze
- Romania (22):
  - Anthos Investigative Site 9022, Baloteşti
  - Anthos Investigative Site 9028, Brasov
  - Anthos Investigative Site 9001, Brăila
  - Anthos Investigative Site 9023, Bucharest
  - Anthos Investigative Site 9019, Bucharest
  - Anthos Investigative Site 9031, Bucharest
  - Anthos Investigative Site 9024, Cluj-Napoca
  - Anthos Investigative Site 9017, Craiova
  - Anthos Investigative Site 9006, Craiova
  - Anthos Investigative Site 9010, Oradea
  - Anthos Investigative Site 9025, Piteşti
  - Anthos Investigative Site 9014, Piteşti
  - Anthos Investigative Site 9012, Satu Mare
  - Anthos Investigative Site 9003, Târgu Mureş
  - Anthos Investigative Site 9004, Târgu Mureş
  - Anthos Investigative Site 9016, Târgu Mureş
  - Anthos Investigative Site 9021, Târgu Mureş
  - Anthos Investigative Site 9007, Timișoara
  - Anthos Investigative Site 9005, Timișoara
  - Anthos Investigative Site 9018, Timișoara
  - Anthos Investigative Site 9013, Timișoara
  - Anthos Investigative Site 9008, Timișoara
- Serbia (12):
  - Anthos Investigative Site 2901, Belgrade
  - Anthos Investigative Site 2903, Belgrade
  - Anthos Investigative Site 2905, Belgrade
  - Anthos Investigative Site 2908, Belgrade
  - Anthos Investigative Site 2911, Belgrade
  - Anthos Investigative Site 2909, Belgrade
  - Anthos Investigative Site 2904, Kragujevac
  - Anthos Investigative Site 2912, Niš
  - Anthos Investigative Site 2910, Novi Pazar
  - Anthos Investigative Site 2906, Smederevo
  - Anthos Investigative Site 2902, Užice
  - Anthos Investigative Site 2907, Zaječar
- Slovakia (7):
  - Anthos Investigative Site 2801, Bardejov
  - Anthos Investigative Site 2807, Bratislava
  - Anthos Investigative Site 2805, Košice
  - Anthos Investigative Site 2806, Lučenec
  - Anthos Investigative Site 2809, Nové Zámky
  - Anthos Investigative Site 2802, Piešťany
  - Anthos Investigative Site 2804, Žilina
- South Africa (10):
  - Anthos Investigative Site 2411, Bellville
  - Anthos Investigative Site 2409, Benoni
  - Anthos Investigative Site 2417, Cape Town
  - Anthos Investigative Site 2408, Centurion
  - Anthos Investigative Site 2412, Durban
  - Anthos Investigative Site 2416, Johannesburg
  - Anthos Investigative Site 2402, Pretoria
  - Anthos Investigative Site 2414, Pretoria
  - Anthos Investigative Site 2415, Somerset West
  - Anthos Investigative Site 2405, Tongaat
- South Korea (17):
  - Anthos Investigative Site 2609, Anyang-si
  - Anthos Investigative Site 2610, Busan
  - Anthos Investigative Site 2606, Busan
  - Anthos Investigative Site 2614, Daegu
  - Anthos Investigative Site 2613, Daejeon
  - Anthos Investigative Site 2615, Goyang-si
  - Anthos Investigative Site 2602, Gwangju
  - Anthos Investigative Site 2611, Gyeonggi-do
  - Anthos Investigative Site 2604, Seongnam-si
  - Anthos Investigative Site 2608, Seoul
  - Anthos Investigative Site 2617, Seoul
  - Anthos Investigative Site 2603, Seoul
  - Anthos Investigative Site 2601, Seoul
  - Anthos Investigative Site 2612, Seoul
  - Anthos Investigative Site 2616, Seoul
  - Anthos Investigative Site 2607, Ulsan
  - Anthos Investigative Site 2605, Yongin-si
- Spain (23):
  - Anthos Investigative Site 1108, A Coruña
  - Anthos Investigative Site 1116, Almería
  - Anthos Investigative Site 1121, Barcelona
  - Anthos Investigative Site 1124, Barcelona
  - Anthos Investigative Site 1120, Barcelona
  - Anthos Investigative Site 1109, Cabra
  - Anthos Investigative Site 1103, Granada
  - Anthos Investigative Site 1111, Jaén
  - Anthos Investigative Site 1118, León
  - Anthos Investigative Site 1104, Madrid
  - Anthos Investigative Site 1117, Madrid
  - Anthos Investigative Site 1106, Madrid
  - Anthos Investigative Site 1113, Madrid
  - Anthos Investigative Site 1105, Málaga
  - Anthos Investigative Site 1110, Murcia
  - Anthos Investigative Site 1115, Oviedo
  - Anthos Investigative Site 1123, Sabadell
  - Anthos Investigative Site 1107, Santiago de Compostela
  - Anthos Investigative Site 1102, Seville
  - Anthos Investigative Site 1122, Seville
  - Anthos Investigative Site 1112, Terrassa
  - Anthos Investigative Site 1101, Valencia
  - Anthos Investigative Site 1119, Vigo
- Sweden (4):
  - Anthos Investigative Site 3303, Danderyd
  - Anthos Investigative Site 3302, Örebro
  - Anthos Investigative Site 3301, Stockholm
  - Anthos Investigative Site 3303, Stockholm
- Turkey (Türkiye) (8):
  - Anthos Investigative Site 3203, Ankara
  - Anthos Investigative Site 3207, Antalya
  - Anthos Investigative Site 3201, Bursa
  - Anthos Investigative Site 3208, Diyarbakır
  - Anthos Investigative Site 3209, Istanbul
  - Anthos Investigative Site 3202, Kayseri
  - Anthos Investigative Site 3206, Mersin
  - Anthos Investigative Site 3204, Samsun
- United Kingdom (25):
  - Anthos Investigative Site 1303, Corby
  - Anthos Investigative Site 1313, Glasgow
  - Anthos Investigative Site 1320, Glasgow
  - Anthos Investigative Site 1315, Hayle
  - Anthos Investigative Site 1311, High Wycombe
  - Anthos Investigative Site 1301, Isleworth
  - Anthos Investigative Site 1316, Kings Lynn
  - Anthos Investigative Site 1324, Lancaster
  - Anthos Investigative Site 1322, Larbert
  - Anthos Investigative Site 1309, Leeds
  - Anthos Investigative Site 1325, Liverpool
  - Anthos Investigative Site 1314, London
  - Anthos Investigative Site 1319, London
  - Anthos Investigative Site 1326, London
  - Anthos Investigative Site 1308, London
  - Anthos Investigative Site 1323, Luton
  - Anthos Investigative Site 1312, Manchester
  - Anthos Investigative Site 1307, Newcastle upon Tyne
  - Anthos Investigative Site 1318, Norwich
  - Anthos Investigative Site 1305, Peterborough
  - Anthos Investigative Site 1321, Romford
  - Anthos Investigative Site 1302, Stevenage
  - Anthos Investigative Site 1310, Stockton-on-Tees
  - Anthos Investigative Site 1317, Stoke-on-Trent
  - Anthos Investigative Site 1306, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com